CLINICAL TRIAL: NCT00129051
Title: Helical Tomotherapy as a Radiotherapy Technique for Treating Pelvic and Abdominal Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA-15-0005
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2005-11

CONDITIONS: Neoplasm Metastasis; Carcinoma
Keywords: tomotherapy; metastatic carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: Tomotherapy

SUMMARY:
Radiation treatment is often used to treat cancer that has spread to the abdomen. It can be very effective at relieving symptoms such as pain, but the radiotherapy itself can cause side-effects such as cramping and diarrhea. This study will investigate whether it is possible to reduce the unwanted side-effects of radiotherapy with a new technology called "helical tomotherapy". Tomotherapy is a new way to deliver radiation in a much more accurate fashion than is currently done, and with less radiation being delivered to normal tissues around the tumor. This study will involve the treatment of 20 patients, who have a spread of their cancer within the abdomen and pelvis, using helical tomotherapy. The dose and energy of radiation will be the same as is currently used - only the delivery system is different. The purpose is to assure that tomotherapy is a safe way to deliver radiation treatment and to investigate whether it will reduce the toxicity of radiation treatment in these patients. Patients will be treated in groups of three until all 20 have been treated. The toxicity of treatment will be measured with a questionnaire for each one. If any unexpected severe treatment complications occur, further accrual will stop.

DETAILED DESCRIPTION:
Radiotherapy is an effective treatment for treating metastatic disease. When used to treat disease in the lower abdomen or pelvis, however, it is frequently associated with gastrointestinal toxicity. The most common symptoms of radiation enteritis are diarrhea, bloating, and abdominal cramping. They are caused by irritation and inflammation of the bowel mucosa, and although the pathophysiology is poorly understood, it is thought to be due in part to malabsorption of bile salts and lactose, imbalances in bacterial flora, disturbances in motility. The true incidence of clinically significant enteritis is not well known and probably underestimated, because the majority of patients with symptoms do not seek medical advice, but is approximately 80% in patients receiving pelvic radiotherapy for gynecologic and rectal tumors. Different approaches have been taken to try to minimize acute small and large bowel toxicity from radiotherapy. Medical management with opioid derivatives, such as loperamide, is often effective for mild cases. Other medications, which try to inhibit the biochemical pathways leading to symptomatic gastroenteritis, have undergone clinical testing with some success. The other approach to minimizing toxicity is to minimize the volume and/or dose of radiation delivered to the small bowel. Simple mechanical devices, such as the "belly board" or a mesh sling, have had some success. With new techniques in intensity-modulated radiotherapy, it may be possible to avoid much of the bowel, or significantly reduce the dose delivered to the bowel, without mechanical intervention or compromising tumour doses. The aim of this trial is to test whether a new and highly sophisticated form of intensity modulated radiotherapy called helical tomotherapy can safely be used to deliver radiotherapy to the abdomen and pelvis. It will also establish whether this treatment modality will allow a reduction in the radiation dose to normal structures and the incidence of radiation-induced bowel injury. Helical tomotherapy is a new form of radiation treatment delivery which will be introduced at the Cross Cancer Institute in late 2001 or early 2002. Unlike standard radiotherapy, in which treatment is delivered through one or a few separate beams, helical tomotherapy delivers treatment with a rotating, intensity-modulated fan beam. The patient is translated through the ring of the gantry while the beam is rotated around, so that the treatment beam forms a helical shape in a similar manner to that of computed tomography (CT) scans. The ring gantry provides a stable platform to perform tomographic verification of both setup and delivered dose. Helical tomotherapy is similar to the NOMOS PeacockTM system currently in clinical use. The PeacockTM system also uses an intensity-modulated fan beam, but because it is an attachment to a standard C-arm linear accelerator, it delivers treatment by a "translate then rotate" method rather than a continuous spiral delivery. Because of the complete freedom of helical tomotherapy to deliver treatment from all angles around the patient and with intensity modulation and inverse treatment planning, it is possible to treat highly complex and irregular target volumes while giving a low radiation dose to surrounding normal structures. This study, along with a parallel study involving the treatment of bone metastases, will involve the first patients to be treated with helical tomotherapy at the Cross Cancer Institute. It will be an important first step in understanding the processes and capabilities of helical tomotherapy in delivering accurate image-guided therapy. It is designed to provide the framework for the next generation of clinical trials using helical tomotherapy in the adjuvant and radical setting. The objectives of the study are as follows:

* To assess whether is is feasible to deliver daily fractionated radiotherapy with helical tomotherapy;
* To assess the acute toxicity associated with the treatment of pelvic and abdominal metastases with helical tomotherapy;
* To test the accuracy of the daily setup verification process inherent in the helical tomotherapy system;
* To perform in vivo dosimetry, where possible;
* To analyze the dose distributions possible with helical tomotherapy planning, and compare to plans obtained using conventional linear accelerator systems.

To accomplish these objectives, the investigators will recruit 20 patients for treatment with helical tomotherapy. Patients with solid malignancy of any primary site with proven or suspected metastatic disease involving the abdomen, pelvis, or bones of the lumbar spine or pelvis will be eligible, provided they are over 18 years of age; signed informed consent is obtained; and there are no contraindications for radiotherapy. The investigators will select patients for enrollment who have a high likelihood (>50%) of suffering from grade 2 or higher acute GI toxicity if standard radiotherapy techniques were used. Treatment will be delivered with the helical tomotherapy system, with the dose plan designed to treat the target volume to a homogeneous dose, while minimizing dose to normal structures including the small bowel. The first 10 patients will be treated with a dose of 2500 cGy in 10 fractions, and the second cohort of 10 patients to 3000 cGy in 10 fractions. The slightly lower than normal dose used for the first cohort is designed to provide an extra margin of safety.

Statistical Considerations: With the doses of radiation used in the current study, the risk of grade 4-5 toxicity using standard treatment techniques is very low. The investigators will, therefore, use observed grade 4-5 acute toxicity as an early stopping rule to monitor the safety of helical tomotherapy. Patients will be accrued onto treatment sequentially, with no more than 3 patients on treatment or within 1 week of completing treatment at any time. If a patient develops a grade 4 toxicity during or shortly after treatment, further accrual will be suspended until such time as the cause of the severe treatment toxicity can be established, and it is determined that treatment to subsequent patients can proceed safely. If a second severe toxicity is observed the trial will close to accrual. For the purposes of the study the risk of grade 4-5 radiation enteritis (using standard radiotherapy techniques) is assumed to be 2% or less. Thus the probability of stopping accrual before trial completion is 0.16 if there is no reduction in toxicity rate with helical tomotherapy (according to binomial probabilities). If the true rate is 1% then the probability of rejecting treatment is 0.01. The acute side effects of treatment will be monitored with the use of a patient symptom questionnaire and physician assessment with history and physical examination. These will be performed pre-treatment, weekly during treatment, and at 1 and 4 weeks post treatment. A secondary endpoint of the study is to test the setup verification process of the helical tomotherapy system. It is designed to automatically detect whether patients are set up accurately for treatment, and to adjust the treatment for day-to-day changes in patient position. For the first 10 patients, the investigators will compare the tomotherapy-derived setup error to the error manually computed by studying the CT image sets. If the computer derived setup error is accurate when compared to the manual evaluation (within 5 mm for at least 80% of measurements), then the automated setup verification process will be utilized for the second cohort of 10 patients. It is estimated that this study will take 3-6 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* Intra-abdominal metastatic cancer

Exclusion Criteria:

* Prior abdominal radiotherapy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-08; Study Completion 2005-11

PRIMARY OUTCOMES:
feasibility and tolerance

SECONDARY OUTCOMES:
efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearcey, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada